CLINICAL TRIAL: NCT00478712
Title: Genetic Analysis of Hirschsprung Disease
Brief Title: Hirschsprung Disease Genetic Study
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 17-01813
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprung
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Study volunteers are asked to provide blood or cheek swab/saliva samples. DNA is extracted from the samples for use in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Families with Hirschsprung Disease: Individuals with Hirschsprung disease and their affected and unaffected relatives.
  Interventions: Other: Identification of genetic causes of Hirschsprung Disease

INTERVENTIONS:
Other: Identification of genetic causes of Hirschsprung Disease — Blood, saliva, or DNA samples are requested from all study participants. The blood or saliva samples are used to isolate DNA in all participants. Blood samples are also used to establish cell lines in some participants.

SUMMARY:
Hirschsprung disease is a genetic condition caused by lack of nerve cells in varying lengths of the intestines. This study will investigate the complex genetic basis of the disease, which involves multiple interacting genetic factors.

DETAILED DESCRIPTION:
Hirschsprung disease (HSCR) is a birth defect resulting from the absence of nerve (ganglion) cells in the gastrointestinal tract. Hirschsprung disease has a population incidence of 1/5000 live births and most often occurs as an isolated condition. However, approximately 30% of HSCR cases are associated with other birth defects such as Down syndrome, deafness, hypopigmentation, and congenital central hypoventilation syndrome. Hirschsprung disease is a genetic condition with autosomal dominant, autosomal recessive, and multigenic patterns of inheritance described.

Dr. Aravinda Chakravarti's laboratory has been investigating the genetics of Hirschsprung disease (HSCR) for more than twenty five years. The goal of this research study is to identify genes harboring causative HSCR mutations and to better understand the complex inheritance of HSCR in families by whole genome mapping and sequencing studies. Specifically, the study aims to determine the frequency with which mutations in any human gene lead to familial and isolated forms of HSCR. Further, the study will collect clinical information and investigate possible genotype - phenotype correlations.

Molecular analysis using markers and sequencing, and statistical analysis of these data will be used to identify regions of human chromosomes where putative HSCR disease genes may be located. In addition, the DNA sequence of known and/or suspected HSCR genes will be assessed in individual patients and their family members, in search of causative HSCR susceptibility variants and variants that may affect presentation of the disease and treatment outcomes. Phenotypic information will include pathology, surgical, and other clinical outcomes related to Hirschsprung disease. This study will hopefully lead to a better understanding of the genetics of HSCR and, further down the road, improved diagnosis, treatment, and genetic counseling.

This study asks volunteers to:

1. Complete a medical/family history questionnaire
2. Provide access to some medical records
3. Submit blood samples from the individual(s) affected with Hirschsprung disease and his/her parents (if available)

ELIGIBILITY:
Inclusion Criteria:

- Individuals with Hirschsprung disease and their first degree relatives (any segment length of disease, with or without other congenital anomalies or health problems, single or multiple affected individuals in family)

Exclusion Criteria:

* Unable or unwilling to provide sample for genetic studies
* Individual, parent, or guardian unable to comprehend and provide informed consent

Ages: 1 Week to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes individuals with Hirschsprung disease and their family members.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2001-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Discovery and characterization of common genetic variation associated with Hirschsprung disease | DNA is isolated up to 1 year after enrollment
  Genome-wide assays of common genetic variation will be assessed using single nucleotide polymorphism (SNP) arrays
Discovery and characterization of copy number variants associated with Hirschsprung disease | DNA is isolated up to 1 year after enrollment
  Copy number variation will be detected using next generation sequencing data and high resolution microarrays that allow for detection of copy number variants across the genome
Discovery and characterization of rare genetic variation associated with Hirschsprung disease | DNA is isolated up to 1 year after enrollment
  Exome sequencing will be used to detect rare variation across all genes in the genome

SECONDARY OUTCOMES:
Correlation of genetic variants with location of transition zone in Hirschsprung disease | Baseline pathology data is obtained up to 1 year after enrollment
  Pathology records and surgical records will be used to determine transition zone
Correlation of genetic variants with risk for enterocolitis in Hirschsprung disease | Baseline clinical data is obtained up to 1 year after enrollment
Characterization of Hirschsprung disease that co-occurs with a known chromosomal disorder | Baseline clinical data is obtained up to 1 year after enrollment
Characterization of Hirschsprung disease that co-occurs with a known single gene syndrome | Baseline clinical data is obtained up to 1 year after enrollment
Characterization of Hirschsprung disease that co-occurs with other congenital anomalies without a known diagnosis | Baseline clinical data is obtained up to 1 year after enrollment
Correlation of genetic variants with need for repeat pull-through surgery in Hirschsprung disease | Baseline clinical data is obtained up to 1 year after enrollment and follow up data is obtained up to 100 years after enrollment
  Assessment of complications that lead to eventual repeat pull-through surgery
Correlation of genetic variants with difficulty controlling stools after pull-through surgery | Baseline clinical data is obtained up to 1 year after enrollment and follow up data is obtained up to 100 years after enrollment
Correlation of genetic variants with chronic constipation after pull-through surgery | Baseline clinical data is obtained up to 1 year after enrollment and follow up data is obtained up to 100 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Aravinda Chakravarti, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Badner JA, Sieber WK, Garver KL, Chakravarti A. A genetic study of Hirschsprung disease. Am J Hum Genet. 1990 Mar;46(3):568-80. PMID 2309705
- [Result] Emison ES, McCallion AS, Kashuk CS, Bush RT, Grice E, Lin S, Portnoy ME, Cutler DJ, Green ED, Chakravarti A. A common sex-dependent mutation in a RET enhancer underlies Hirschsprung disease risk. Nature. 2005 Apr 14;434(7035):857-63. doi: 10.1038/nature03467. PMID 15829955
- [Result] Gabriel SB, Salomon R, Pelet A, Angrist M, Amiel J, Fornage M, Attie-Bitach T, Olson JM, Hofstra R, Buys C, Steffann J, Munnich A, Lyonnet S, Chakravarti A. Segregation at three loci explains familial and population risk in Hirschsprung disease. Nat Genet. 2002 May;31(1):89-93. doi: 10.1038/ng868. Epub 2002 Apr 15. PMID 11953745
- [Result] Arnold S, Pelet A, Amiel J, Borrego S, Hofstra R, Tam P, Ceccherini I, Lyonnet S, Sherman S, Chakravarti A. Interaction between a chromosome 10 RET enhancer and chromosome 21 in the Down syndrome-Hirschsprung disease association. Hum Mutat. 2009 May;30(5):771-5. doi: 10.1002/humu.20944. PMID 19306335
- [Result] Emison ES, Garcia-Barcelo M, Grice EA, Lantieri F, Amiel J, Burzynski G, Fernandez RM, Hao L, Kashuk C, West K, Miao X, Tam PK, Griseri P, Ceccherini I, Pelet A, Jannot AS, de Pontual L, Henrion-Caude A, Lyonnet S, Verheij JB, Hofstra RM, Antinolo G, Borrego S, McCallion AS, Chakravarti A. Differential contributions of rare and common, coding and noncoding Ret mutations to multifactorial Hirschsprung disease liability. Am J Hum Genet. 2010 Jul 9;87(1):60-74. doi: 10.1016/j.ajhg.2010.06.007. PMID 20598273
- [Result] Kapoor A, Jiang Q, Chatterjee S, Chakraborty P, Sosa MX, Berrios C, Chakravarti A. Population variation in total genetic risk of Hirschsprung disease from common RET, SEMA3 and NRG1 susceptibility polymorphisms. Hum Mol Genet. 2015 May 15;24(10):2997-3003. doi: 10.1093/hmg/ddv051. Epub 2015 Feb 9. PMID 25666438
- [Result] Chatterjee S, Kapoor A, Akiyama JA, Auer DR, Lee D, Gabriel S, Berrios C, Pennacchio LA, Chakravarti A. Enhancer Variants Synergistically Drive Dysfunction of a Gene Regulatory Network In Hirschsprung Disease. Cell. 2016 Oct 6;167(2):355-368.e10. doi: 10.1016/j.cell.2016.09.005. Epub 2016 Sep 29. PMID 27693352
- See also: Chakravarti, Johns Hopkins Medical Institution (JHMI) Faculty Biography Page — https://igm.jhmi.edu/faculty/aravinda-chakravarti